CLINICAL TRIAL: NCT03851575
Title: Accelerated Treatment of Endocarditis
Acronym: POETII
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Herlev Hospital (Other); Nordsjaellands Hospital (Other); Zealand University Hospital (Other); Odense University Hospital (Other); Aarhus University Hospital (Other); Lund University Hospital (Other)
Responsible Party: Principal Investigator, Kasper Iversen, Associate professor, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-18028566
Record Dates: First submitted 2018-12-03; First posted 2019-02-22 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Infectious Endocarditis
MeSH Terms: conditions — Endocarditis, Subacute Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (Active Comparator): Usual guideline therapy
  Interventions: Other: Usual guideline therapy
- Accelerated arm (Experimental): Accelerated treatment of endocarditis
  Interventions: Other: Accelerated treatment of endocarditis

INTERVENTIONS:
Other: Accelerated treatment of endocarditis — For the three main bacteria species we shorten the duration of antibiotic treatment
  Arms: Accelerated arm
Other: Usual guideline therapy — Usual guideline therapy
  Arms: Control arm

SUMMARY:
Existing guidelines recommend a duration of antibiotic treatment of endocarditis of 4-6 weeks with one or two types of intravenously administered antibiotics. The long hospitalization increases several risks for the patient, including mental strain and increased loss of function. Furthermore, it poses a significant burden on health systems. Current guidelines fail to use available data collected from patients (echo, temperature, CRP, leukocytes, procalcitonin etc.) to determine duration of treatment. A strategy including these data in treatment algorithms ensures an individualized treatment, targeting the patient's course and response to treatment. Thus, the purpose of this open-label, prospective, non-inferiority, RCT study is to investigate the safety and effectiveness of shortening treatment of endocarditis based on the individual patient's initial treatment response, sampling 750 patients, approx. 200 patients with each type of bacteria (Streptococci; Enterococcus faecalis; Staphylococcus aureus). Interim analysis will be conducted when 150 patients have been included, to assess the frequency of the event rate and inclusion rate in order to adjust the intended size of the study population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients hospitalized and diagnosed with bacterial, left-sided endocarditis as determined by the department clinician responsible based on the revised Duke criteria.
2. The patient may be included <14 days after beginning of relevant antibiotic treatment.
3. Left-sided endocarditis with one of the following microorganisms: Streptococci; Enterococcus faecalis; Staphylococcus aureus.
4. Patients ≥ 18 years.

Exclusion Criteria:

1. Known / suspected immunocompetence (HIV, chemotherapy, prednisolone treatment (> 20 mg / day)).
2. Incapability to give informed consent for participation.
3. Relapse Endocarditis (Endocarditis with the same bacteria within six months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2019-01-17 (Actual); Primary Completion 2023-06-10 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
Primary composite endpoint | 6 monts after randomization
  Number of patients with at least one of the following: Death (yes/no); Embolisms (yes/no); Bacteraemia with the same microorganism (yes/no), surgery not planned at randomization (yes/no).

SECONDARY OUTCOMES:
Quality of life | 6 monts after randomization and after
  Quality of life assessed by completing short version 36 (SF 36) version 2
Expenses | 6 monts after randomization
  Expenses associated with hospitalization and treatment of the disease. I.E., expenses to admission, examinations and medicine
Duration of hospitalization | 6 monts after randomization
  Duration of hospitalization
Death | 6 monts after randomization
  Number of patients that die
Embolisms | 6 monts after randomization
  Number of patients that have an embolism
Bacteraemia with the same microorganism, | 6 monts after randomization
  Number of patients that have Bacteraemia with the same microorganism
Surgery not planned at randomization | 6 monts after randomization
  Number of patients that have Surgery not planned at randomization

CONTACTS AND LOCATIONS:
Overall Officials: Henning Bundgaard, MD, Study Chair — Rigshospitalet, Denmark
Locations (7):
- Denmark (7):
  - Skejby Sygehus, Aarhus
  - Rigshospitalet, Copenhagen
  - Gentofte Hospital, Copenhagen
  - Herlev Hoslpital, Copenhagen
  - Hillerød Hospital, Hillerød
  - Odense Sygehus, Odense
  - Roskilde Sygehus, Roskilde

IPD SHARING:
Plan to Share IPD: Undecided